CLINICAL TRIAL: NCT02636894
Title: Evaluation of the Efficacy of Restylane Silk in the Treatment of Cheek Fold (Radial Smile Lines)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amanda D. Spear, CCRC (Other)
Responsible Party: Sponsor-Investigator, Amanda D. Spear, CCRC, Brian Biesman, MD, Nashville Centre for Laser and Facial Surgery
Organization: Nashville Centre for Laser and Facial Surgery (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Restylane Silk
Record Dates: First submitted 2015-12-16; First posted 2015-12-22 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Smile Lines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Restylane Silk (Other): Restylane Silk
  Interventions: Device: Restylane Silk

INTERVENTIONS:
Device: Restylane Silk

SUMMARY:
Filler study for smile lines in cheek folds

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 21-65 years of age
* Willing to comply with study visits and procedures
* Willingness to refrain form surgical, laser, or injectable treatments in cheek region during study

Exclusion Criteria:

* History of trauma, acne scarring, burns, or other changes to skin in treatment area
* Use of botulinum toxin in the lateral cheeks/perioral region in past 6 months
* Use of injectable fillers in the lateral cheeks/perioral within last 2 years
* History of facelift in the last year
* History of facial nerve palsy

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Evaluation of the Efficacy of Restylane Silk in the Treatment of Cheek folds (Radial Smile Lines) | 6 months
  Improvement of subjects based on 5 point global aesthetic scale (GAIS)

IPD SHARING:
Plan to Share IPD: No